CLINICAL TRIAL: NCT04760093
Title: A Multicenter Pilot Study to Evaluate the Effect of EVOO on Lipid Parameters
Acronym: EVOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ralph Hamill (Other)
Responsible Party: Sponsor-Investigator, Ralph Hamill, Cardiologist, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1639676
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases
Keywords: Lipoproteins, HDL; Extra virgin olive oil
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: In this study, subjects will be randomized to one of two research arms. Subjects in the first research arm will be given low polyphenol concentration EVOO, followed by high polyphenol concentration EVOO for consumption. Subjects in the second research arm will be given high polyphenol concentration EVOO, followed by low polyphenol concentration EVOO for consumption. There will be a 14- day washout period in between administration of either low or high polyphenol concentration EVOO.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pharmacists will assign participants to one of the research arms following a randomization schedule, and will maintain a study log not accessible to the investigators or care provider. Study coordinators will remain blinded when distributing the bottles of EVOO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-to-High group (Other): As this is a crossover study, each participant will be assigned to each treatment intervention. Participants (randomly) assigned to Arm 1 will first receive low polyphenol concentration EVOO for consumption, followed by high polyphenol concentration EVOO for consumption following a 14- day washout phase.
  Interventions: Dietary Supplement: Low polyphenol concentration extra virgin olive oil (EVOO); Dietary Supplement: High polyphenol concentration extra virgin olive oil (EVOO)
- High-to-Low group (Other): As this is a crossover study, each participant will be assigned to each treatment intervention. Participants (randomly) assigned to Arm 2 will first receive high polyphenol concentration EVOO for consumption, followed by low polyphenol concentration EVOO for consumption following a 14- day washout phase.
  Interventions: Dietary Supplement: Low polyphenol concentration extra virgin olive oil (EVOO); Dietary Supplement: High polyphenol concentration extra virgin olive oil (EVOO)

INTERVENTIONS:
Dietary Supplement: Low polyphenol concentration extra virgin olive oil (EVOO) — Subjects will complete a consecutive 28-day period of consuming low polyphenol concentration EVOO daily.
Dietary Supplement: High polyphenol concentration extra virgin olive oil (EVOO) — Subjects will complete a consecutive 28-day period of consuming high polyphenol concentration EVOO daily.

SUMMARY:
The purpose of this multi-center, double-blinded pilot study is to determine if extra virgin olive oil (EVOO) has a positive effect on HDL cholesterol levels and anti-inflammatory markers for subjects diagnosed with cardiovascular disease (CVD) and to determine if the polyphenol concentration is proportional to those effects. Subjects will complete consecutive 28-day periods (with a 14-day washout between) in which they will either consume the low polyphenol concentration EVOO daily or the high polyphenol concentration EVOO. In a double-blinded manner, each subject will be his or her own control with a 14-day washout between study periods. HDL levels and other parameters will be measured after each period of the protocol. The investigators anticipate HDL levels will improve with both olive oils. The investigators expect the high polyphenol concentration EVOO will show a greater effect than the EVOO with a low polyphenol concentration. EVOO with high polyphenol concentration may be a simple method to reduce the risk of secondary CVD events.

DETAILED DESCRIPTION:
Study Design:

A multi-center, double-blinded pilot study to determine if extra virgin olive oil (EVOO) has a positive effect on HDL cholesterol levels and anti-inflammatory markers for subjects diagnosed with cardiovascular disease (CVD) and to determine if the polyphenol concentration is proportional to those effects. Subjects will complete consecutive 28-day periods (with a 14-day washout between) in which they will either consume the low polyphenol concentration EVOO daily or the high polyphenol concentration EVOO. In a double-blinded manner, each subject will be his or her own control with a 14-day washout between study periods.

Hypothesis:

Subjects will demonstrate greater improvements in HDL cholesterol levels, other lipid parameters, and inflammatory markers by adding EVOO to their diets. Consumption of EVOO with high polyphenol concentration will improve these parameters more than consumption of EVOO with low polyphenol concentration.

Specific Aims:

1. To determine if daily consumption of EVOO will increase HDL cholesterol levels after 28 days.
2. To determine if daily consumption of high polyphenol concentration EVOO increases HDL cholesterol levels more than EVOO with a low polyphenol concentration (same dosing).
3. To determine the feasibility of this type of study and the possibility of a larger study over a longer time period.

Study Methods:

Prior to enrolling subjects, the study staff will order a generic brand EVOO through the hospital nutritional services department. At the same time, EVOO with a reported high polyphenol concentration will be ordered from a local olive oil specialty store.

Olive oil testing: Eurofins Microbiology Laboratories, Inc. will test a sample of each batch of olive oil for polyphenol concentration prior to dispensing. The method is based on direct extraction of the biophenolic minor polar compounds from olive oil by means of a methanol solution and subsequent quantification by HPLC-MS/MS. Commercially available polyphenol standards are used to identify and quantify individual phenolic compounds, focusing on those most abundant in olive oils.

Study subject blood testing: Approximately 20 ml of blood will be obtained at five different study visits for a total of 100 ml of blood over 12 weeks.

Baseline serum and plasma blood samples will be taken prior to olive oil supplementation. Follow-up blood samples will be taken at four other times points.

Serum total lipid profiles will be evaluated in the mass spectrometry core at the Maine Medical Center Research Institute (MMCRI). Additionally, inflammatory markers, including CRP, IL-6 and TNFalpha, will be determined by enzyme-linked immunosorbent assay (ELISA). Serum will be prepared by collecting 10 ml of blood into red cap tubes. Blood will be allowed to coagulate for 15-20 minutes at room temperature and then centrifuged at 1500 - 2000g, and the supernatant pipetted off and stored frozen at -65ºC. Plasma samples will be prepared from 6 ml of blood collected into 10 ml ACD (Acid Citrate Dextrose) anticoagulant tubes and processed within 1h. The white blood cell fraction will be prepared by centrifugation at 1,500-2000g for 15 minutes. The middle layer of white cells will be pipetted off and stored frozen at -60ºC. The investigators will determine the lipidomic profiles of white blood cells as well as caveolin-1 protein levels.

Lipid panels, which test total cholesterol, HDL, LDL, and triglycerides, will be run on remaining blood samples at the local laboratory. All blood testing- associated costs will be paid for with study funds from the MaineHealth Cardiology Service Line.

Other study measures: Vital signs including body weight, blood pressure and heart rate will be measured at each visit.

Subjects will maintain a study diary documenting each dose of EVOO. They will be asked to measure out 1 ounce of olive oil in a cup given to them by the study team, and consume it with bread, in a smoothie, or by drinking it plain. Compliance with EVOO consumption will be calculated from the diary (%). Study compliance will also be measured by ounces of product returned (%). Subjects receive 30 ounces of EVOO to cover 28 days, therefore, 2 ounces of returned olive oil after each study arm will be counted as 100% compliance.

Sample Size Considerations:

As this is a pilot study, the investigators utilized data available in the literature to estimate sample size. A study evaluating the effect of HDL on older age life expectancy reported a mean HDL of 47.5 with a standard deviation of 12.1 among subjects who lived to be older than 85 years. Using this estimate, and anticipating to find a 3 point difference in HDL among the two study groups, the investigators need to recruit 276 participants. However, as this is a pilot study and the investigators have limited funding, they will start by recruiting 90 subjects. With additional funding secured from a grant in the future, the study could be expanded in order to achieve the desired power of 80%.

Data Analysis:

For the purpose of this study, the investigators will attempt to detect differences in HDL and other biomarkers of cardiovascular health in subjects who consumed both low polyphenol concentration vs. high polyphenol concentration EVOO. Medical record numbers will not be included in the dataset for analysis. Descriptive statistics will be used to summarize the demographic and clinical characteristics of subjects included in the study, with continuous variables presented as a mean +- standard deviation and categorical variables as frequencies/percentages of the total. Student t tests and chi-squared tests will be conducted to compare data between the low vs. high polyphenol EVOO groups. A time series plot will be generated in order to demonstrate the change in HDL over time by level of polyphenol consumed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Both males and females will be included
* Known cardiovascular disease as documented by ICD code
* HDL < 40 documented within the past 12 months
* Able to fast for 12 hours prior to blood draws

Exclusion Criteria:

* Unwilling or unable to provide informed consent for any reason
* Inability to adhere to protocol for any reason
* Currently using EVOO on a daily basis
* Change in use of lipid lowering medications or supplements in the past 90 days or plans to change during study participation
* HDL > 40 on baseline blood draw
* Significant change in diet or exercise in the past 30 days or plan to do so during the study time period
* Allergic to olive oil
* Unable to fast for 12 hours prior to blood draws
* Pregnancy
* Enrolled in another interventional research study
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
HDL | HDL will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in HDL in subjects who consumed low polyphenol vs. high polyphenol EVOO.

SECONDARY OUTCOMES:
IL-6 | IL-6 will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in IL-6 in subjects who consumed low polyphenol vs. high polyphenol EVOO.
CRP | CRP will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in CRP in subjects who consumed low polyphenol vs. high polyphenol EVOO.
Lipid panel | Lipid panels will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in lipid panel results in subjects who consumed low polyphenol vs. high polyphenol EVOO.
Blood pressure | Blood pressure will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in blood pressure in subjects who consumed low polyphenol vs. high polyphenol EVOO.
Heart rate | Heart rate will be measured in each subject within 28 days before and within 28 days after consuming either low or high polyphenol EVOO.
  Average difference in heart rate in subjects who consumed low polyphenol vs. high polyphenol EVOO.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hamill, MD, Principal Investigator — Maine Medical Partners
Locations (3):
- United States (3):
  - Mid Coast Cardiology, Brunswick, Maine
  - Pen Bay Medical Center, Rockport, Maine
  - Maine Medical Partners Cardiology, Scarborough, Maine

IPD SHARING:
Plan to Share IPD: No
Investigators will only share aggregate data from this study with other researchers.

REFERENCES:
- [Background] Buckland G, Travier N, Barricarte A, Ardanaz E, Moreno-Iribas C, Sanchez MJ, Molina-Montes E, Chirlaque MD, Huerta JM, Navarro C, Redondo ML, Amiano P, Dorronsoro M, Larranaga N, Gonzalez CA. Olive oil intake and CHD in the European Prospective Investigation into Cancer and Nutrition Spanish cohort. Br J Nutr. 2012 Dec 14;108(11):2075-82. doi: 10.1017/S000711451200298X. Epub 2012 Sep 25. PMID 23006416
- [Background] Caporaso, N., Savarese, M., Paduano, A., Guidone, G., De Marco, E., & Sacchi, R. (2015). Nutritional quality assessment of extra virgini olive oil from the Italian retail market: Do natural antioxidants satisfy EFSA health claims? Journal of Food Composition and Analysis, 40, 154-162. doi:10.1016/j.jfca.2014.12.012
- [Background] Estruch R, Lamuela-Raventos RM, Ros E. The Bitter Taste of Extra Virgin Olive Oil for a Sweet Long Life. J Am Coll Cardiol. 2020 Apr 21;75(15):1740-1742. doi: 10.1016/j.jacc.2020.02.043. No abstract available. PMID 32299584
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Fiorini D, Boarelli MC, Conti P, Alfei B, Caprioli G, Ricciutelli M, Sagratini G, Fedeli D, Gabbianelli R, Pacetti D. Chemical and sensory differences between high price and low price extra virgin olive oils. Food Res Int. 2018 Mar;105:65-75. doi: 10.1016/j.foodres.2017.11.005. Epub 2017 Nov 6. PMID 29433259
- [Background] Guasch-Ferre M, Liu G, Li Y, Sampson L, Manson JE, Salas-Salvado J, Martinez-Gonzalez MA, Stampfer MJ, Willett WC, Sun Q, Hu FB. Olive Oil Consumption and Cardiovascular Risk in U.S. Adults. J Am Coll Cardiol. 2020 Apr 21;75(15):1729-1739. doi: 10.1016/j.jacc.2020.02.036. Epub 2020 Mar 5. PMID 32147453
- [Background] Khan TM, Iqbal S, Rashid MA. Comparison Of Lipid Lowering Effect Of Extra Virgin Olive Oil And Atorvastatin In Dyslipidaemia In Type 2 Diabetes Mellitus. J Ayub Med Coll Abbottabad. 2017 Jan-Mar;29(1):83-86. PMID 28712181
- [Background] Rahilly-Tierney CR, Spiro A 3rd, Vokonas P, Gaziano JM. Relation between high-density lipoprotein cholesterol and survival to age 85 years in men (from the VA normative aging study). Am J Cardiol. 2011 Apr 15;107(8):1173-7. doi: 10.1016/j.amjcard.2010.12.015. Epub 2011 Feb 4. PMID 21296318
- [Background] Servili M, Esposto S, Fabiani R, Urbani S, Taticchi A, Mariucci F, Selvaggini R, Montedoro GF. Phenolic compounds in olive oil: antioxidant, health and organoleptic activities according to their chemical structure. Inflammopharmacology. 2009 Apr;17(2):76-84. doi: 10.1007/s10787-008-8014-y. PMID 19234678